CLINICAL TRIAL: NCT04373395
Title: A Prospective, Single-arm, Multicenter, Exploratory Study to Evaluate the Efficacy and Safety of D-CLAG Regimen in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Decitabine+Cladribine+Cytarabine+Granulocyte Colony-stimulating Factor (D-CLAG) for Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Zhejiang Provincial People's Hospital (Other); First People's Hospital of Hangzhou (Other); Zhejiang Provincial Tongde Hospital (Other); Jinhua Central Hospital (Other); Huizhou Municipal Central Hospital (Other); The Sixth Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry); Hanhui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, He Huang, President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-CLAG-ZJU
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- D-CLAG (Experimental): Administration of D-CLAG regimen (Decitabine+Cladribine+Cytarabine+Granulocyte Colony Stimulating Factor)
  Interventions: Procedure: D-CLAG

INTERVENTIONS:
Procedure: D-CLAG — Decitabine+Cladribine+Cytarabine+Granulocyte Colony Stimulating Factor

SUMMARY:
A prospective, single-arm, multicenter, exploratory study to evaluate the efficacy and safety of D-CLAG regimen in the treatment of relapsed or refractory acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (non-acute promyelocytic leukemia) must be diagnosed before enrollment. Diagnostic criteria refer to WHO (World Health Organization) classification.
* Refractory or relapsed AML: refractory is defined as the failure of CR after 2 courses of standard induced remission therapy (2 courses of idarubicin+cytarabine (IA) regimen or 1 course of IA regimen + 1 course of high dose cytarabine); Relapse is defined as the blast cells >5% in bone marrow or presence of extramedullary leukemia for patient who achieved CR before.
* Age 18-70.
* Eastern cancer cooperation group (ECOG) ≤2.
* Creatinine clearance ≥30 mL/min (estimated glomerular filtration rate (eGFR) according to the Cockcroft-Gault formula or Modification of Diet in Renal Disease (MDRD) formula).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3× upper limit of normal range (ULN), total bilirubin ≤2×ULN.
* Echocardiography (ECHO) showed left ventricular ejection fraction (LVEF)≥50%.
* Life expectancy >8 weeks.
* Voluntarily sign the informed consent and understand and comply with the requirements of the study.

Exclusion Criteria:

* White blood cell (WBC) > 50 * 109 / L
* Patients who have received salvage treatment with D-CLAG.
* Current active cardiovascular disease, such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease according to the New York heart association (NYHA) functional classification, or a history of myocardial infarction within 6 months prior to screening.
* Other serious diseases that may limit patient participation in the trial (e.g. progressive infections, uncontrolled diabetes).
* Pregnant or nursing women.
* Unable to understand or follow the research protocol or unable to sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | Complete blood count recovery or 1 month after 1 course of D-CLAG regimen
  Complete remission rate after 1 course of D-CLAG regimen

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China